CLINICAL TRIAL: NCT02278679
Title: Validation of the DiRECT Proficiency Tool
Brief Title: Digital Rectal Exam Proficiency Tool
Acronym: DiRECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Tracey Krupski, MD, M.D. Associate Professor of Urology, University of Virginia
Other Study IDs: 17658
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia; Prostate Cancer
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Anesthitized patient: First, it will be validated on 120 anesthetized patients undergoing prostate surgery comparing responses on the digital rectal exam clinical tool (DiRECT) from both expert and novice clinicians, with surgical pathology reports.
  Interventions: Procedure: Digital Rectal Exam
- Standardized patients: During a standardized patient exercise focusing on digital rectal exam in the University of Virginia School of Medicine curriculum, 160 second-year medical students will be given the DiRECT to document their examination. An attending physician will also attend the standardized patient exercise and document their examination for comparison with the medical students.
- Clinic patient: The third phase includes 8 residents and up to10 attendings in the Urology clinic, who will independently complete the DiRECT documenting their DRE in the course of usual care.

INTERVENTIONS:
Procedure: Digital Rectal Exam — The DRE digital rectal exam is an essential component of physical examination, but physicians enter their residency having neither been appropriately exposed nor trained in performing DREs. , the attending physician, resident physician(s), and medical student(s) will each perform a digital rectal exam on the subject, and independently document their examination on the DiRECT instrument.
  Groups: Anesthitized patient

SUMMARY:
A digital rectal exam proficiency tool, titled the 'DiRECT' was developed based on the consensus of 10 experts. The purpose of this study is to validate this tool for use in both undergraduate and graduate medical education .

DETAILED DESCRIPTION:
First, it will be validated on 120 anesthetized patients undergoing prostate surgery, comparing responses on the digital rectal exam clinical tool (DiRECT) from both expert and novice clinicians, with surgical pathology reports. The second phase of validation will involve the participation of standardized patients, medical students and MUTA (medical urology teaching associate). During a standardized patient exercise focusing on digital rectal exam in the University of Virginia School of Medicine curriculum, 160 second-year medical students will be given the DiRECT to document their examination. An attending physician will also attend the standardized patient exercise and document their examination for comparison with the medical students.

The third phase includes 8 residents and up to10 attendings in the Urology clinic, who will independently complete the DiRECT documenting their DRE in the course of usual care.

Comparison of faculty and student/trainee responses in all phases will be used for validation of the clinical tool for further use in medical education.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are patients:

* Patients who are male and adults ≥ 30 years of age
* Standardized patients between the ages of 30-80 years participating in the University of Virginia School of Medicine activity for second-year students learning digital rectal exams

Subjects who are clinicians:

• Attending physician, resident physician, or medical student scrubbed in for a prostatectomy or cystectomy, seeing patients in urology clinic, or participating in the School of Medicine activity for second year students learning digital rectal exams

Exclusion Criteria:

List the criteria for exclusion

* Patients who do not have a prostate
* Patients with previous pelvic/perineal surgery
* Previously enrolled in this study

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Benign Prostate Hypertrophy, Prostate Cancer or routine digital exam being seen by Urology Attendings, residents or medical students.
Sampling Method: Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Validate DiRECT tool | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Krupski, M.D., Principal Investigator — University of Virginia, Dept of Urology; Raymond A Costabile, M.D., Study Chair — University of Virginia, Dept of Urology
Locations (1):
- University of Virginia Health System, Dept of Urology, Charlottesville, Virginia, United States